CLINICAL TRIAL: NCT01827930
Title: Phase III Trial Evaluating the Effectiveness of a Dose Adjustment of IM on the Molecular Response in Patients With LMC in Chronic Phase Treated With IM 400 mg / Day for at Least Two Years, Complete Cytogenetic Response for at Least One Year
Brief Title: Phase III Trial Evaluating the Effectiveness of a Dose Adjustment of Imatinib Mesylate on the Molecular Response
Acronym: MIM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties of enrolment of Patient
Sponsor: Institut Bergonié (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB2009-07; 2008-007094-20 (EudraCT Number)
Record Dates: First submitted 2012-11-05; First posted 2013-04-10 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
Keywords: chronic myeloid leukemia in chronic phase; residual plasma IM concentration; adapted strategy
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; Tablets

STUDY DESIGN:
Intervention Model Description: IM concentration < 1000ng/mL Randomized Cohort : "adapted strategy" versus "standard strategy" / IM concentration >= 1000ng/mL Parallel Cohort: "standard strategy"
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Imatinib 600 (Randomized trial) (Experimental): Randomized Cohort: Adapted strategy of dosage of Imatinib Mesylate : 600mg/d po
  Interventions: Drug: Imatinib Mesylate 600 MG Oral Tablet
- Imatinib 400 (Randomized trial) (Active Comparator): Randomized Cohort: Standard strategy of dosage of Imatinib Mesylate : 400mg/d po
  Interventions: Drug: Imatinib Mesylate 400 MG Oral Tablet
- Imatinib400 (Cohort) (Other): Parallel Cohort: Standard strategy of dosage of Imatinib Mesylate : 400mg/d po
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate 600 MG Oral Tablet — Imatinib Mesylate for CP CML
  Other Names: GLIVEC
  Arms: Imatinib 600 (Randomized trial)
Drug: Imatinib Mesylate 400 MG Oral Tablet — Imatinib Mesylate for CP CML
  Other Names: GLIVEC
  Arms: Imatinib 400 (Randomized trial)
Drug: Imatinib Mesylate — Imatinib Mesylate for CP CML
  Other Names: GLIVEC
  Arms: Imatinib400 (Cohort)

SUMMARY:
The Imatinib Mesylate at a dose of 400 mg / day is the standard treatment for patients with CML-CP. Recent studies show that the quality of response rate (complete cytogenetic response and major molecular response rate) is dependent on the residual plasma Imatinib.

DETAILED DESCRIPTION:
The Imatinib Mesylate at a dose of 400 mg / day is the standard treatment for patients with CML-CP. Recent studies show that the quality of response rate (complete cytogenetic response and major molecular response rate) is dependent on the residual plasma Imatinib. This study aims to evaluate the effectiveness of a strategy for dose adjustment of Imatinib Mesylate based on the measurement of the residual plasma imatinib in patients treated for at least 2 years Imatinib 400 mg / d in complete cytogenetic response for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CML-CP treated for at least two years by Imatinib Mesylate 400 mg / d,
2. Patients in complete cytogenetic response for at least 1 year
3. Patients with residual disease detectable by quantitative RT-PCR (RQ-PCR)
4. ECOG ≤ 2,
5. Age ≥ 18 years
6. Signed informed consent,
7. Membership of a social security system

Exclusion Criteria:

1. Patients with CML-CP Philadelphia chromosome negative diagnosis.
2. Patients previously treated with Imatinib Mesylate at doses above 400 mg / day
3. Patient with non-hematologic toxicity of grade III or IV in Imatinib Mesylate 400mg / d
4. Patient with a medical condition endocrine, psychiatric, neurological, renal, hepatic or cardiac progressive uncontrolled by medical treatment
5. Pregnant or breastfeeding women, women of childbearing potential not using a contraceptive method effective
6. Known HIV positive
7. Patients previously treated with another tyrosine kinase inhibitor
8. Patient participating in another interventional clinical trial
9. History of non-compliance to Imatinib Mesylate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ETIENNE Gabriel, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

REFERENCES:
- See also: Registre des essais cliniques de l'INCa — https://www.e-cancer.fr/Professionnels-de-sante/Le-registre-des-essais-cliniques
- See also: Site internet du promoteur, l'Institut Bergonié — https://www.bergonie.fr/les-essais-cliniques

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Cohort)
Started | 24 | 25 | 19
Completed | 24 | 25 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients included, regardless of whether or not treatment was administered, and regardless violations of any eligibility criteria. This population corresponds to Intention to treat population for randomized study, and population assessable for the primary endpoind for the parralel cohort.
Groups:
- Imatinib400 (Parallel Cohort): Parallel Cohort: Standard strategy of dosage of Imatinib Mesylate : 400mg/d po
  Imatinib Mesylate: Imatinib Mesylate for CP CML
- Total: Total of all reporting groups
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort) | Total
Number analyzed (Participants) | 24 | 25 | 19 | 68
Age, Continuous [Median (Full Range); unit: years] | 50.6 [27.7 to 72.0] | 52.7 [25.1 to 79.1] | 65.3 [34.3 to 80.4] | 54.5 [25.1 to 80.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 6 | 16
  Male | 20 | 19 | 13 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 24 | 25 | 19 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Presenting a Decline of the BCR-ABL Transcript Rate at 12 Months From Baseline - Randomised Study
Description: The BCR-ABL transcript rate was analysed by molecular biology by RQ-PCR at study entry, 3 months, 6 months, 9 months and 12 months.
  Treatment is considered effective at 12 months if:
  * for patients with an inclusion transcript rate less than 0.1%: the transcript rate at 12 months is less or equal to 0.001% or undetectable.
  * for patients with an inclusion transcript rate greater than 0.1% : the transcript rate at 12 months is less or equal to 0.1% or undetectable.
  If BCR-ABL transcript level was unavailable at M12, the treatment was considered ineffective.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 24 | 25 | 19
percentage of patients | 29.2 [12.6 to 51.1] | 32.0 [14.9 to 53.5] | 10.5 [1.3 to 33.1]

2. Secondary Outcome: Rate of Decline of 2-log of the BCR-ABL Transcript Rate at 3 ,6, 9 and 12 Months From Baseline - Randomised Study
Description: The BCR-ABL transcript rate was analysed by molecular biology by RQ-PCR at study entry, 3 months, 6 months, 9 months and 12 months.
  Efficacy was also evaluated at 3, 6, 9 and 12 months in terms of decreasing the rate of BCR-ABL transcripts of 2 logarithms, relative to the initial value (inclusion). The lack of data on the transcript rate was considered as failure (no decrease).
Time Frame: 3, 6, 9 and 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 24 | 25 | 19
percentage of patients
  3 months | 4.2 [0.1 to 21.1] | 0 [NA to NA] — insufficient number of participants with events | 0 [NA to NA] — insufficient number of participants with events
  6 months | 4.2 [0.1 to 21.1] | 0 [NA to NA] — insufficient number of participants with events | 0 [NA to NA] — insufficient number of participants with events
  9 months | 0 [NA to NA] — insufficient number of participants with events | 0 [NA to NA] — insufficient number of participants with events | 0 [NA to NA] — insufficient number of participants with events
  12 months | 4.2 [0.1 to 21.1] | 0 [NA to NA] — insufficient number of participants with events | 0 [NA to NA] — insufficient number of participants with events

3. Secondary Outcome: Molecular Response at 3, 6, 9 and 12 Months
Description: The molecular response is defined by the measurement of BCR-ABL transcript rate by quantitative RT-PCR (RQ-PCR) on peripheral venous blood according to international standards.
  It is defined as:
  * Major Molecular Response (MMR): BRC-ABL transcript rate ≤ 0.1%
  * Complete Molecular Response (CMR): transcript BCR-ABL undetectable and non quantifiable.
Time Frame: 3, 6, 9 and 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of patient
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 24 | 25 | 19
percentage of patient
  3 months - CMR | 12.5 [2.7 to 32.4] | 8.0 [1.0 to 26.0] | 0 [NA to NA] — insufficient number of participants with events
  3 months : MMR | 75.0 [53.3 to 90.2] | 80.0 [59.3 to 93.2] | 78.9 [54.4 to 93.9]
  6 months : CMR | 4.2 [0.1 to 21.1] | 8.0 [1.0 to 26.0] | 0 [NA to NA] — insufficient number of participants with events
  6 months : MMR | 87.5 [67.6 to 97.3] | 72.0 [50.6 to 87.9] | 73.7 [48.8 to 90.9]
  9 months : CMR | 20.8 [7.1 to 42.2] | 4.0 [0.1 to 20.4] | 5.3 [0.1 to 26.0]
  9 months : MMR | 66.7 [44.7 to 84.4] | 68.0 [46.5 to 85.1] | 68.4 [43.4 to 87.4]
  12 months : CMR | 8.3 [1.0 to 27.0] | 4.0 [0.1 to 20.4] | 5.3 [0.1 to 26.0]
  12 months : MMR | 83.3 [62.6 to 95.3] | 76.0 [54.9 to 90.6] | 63.2 [38.4 to 83.7]

4. Secondary Outcome: Time to Complete Molecular Response (CMR) and Major Molecular Response (MMR)
Description: Time to complete molecular response was defined by the time from inclusion/randomization and the first CMR.
Time Frame: From date of randomization until the date of complete molecular response (up to 12 months)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 24 | 25 | 18
months
  CMR: number analyzed (Participants) | 7 | 3 | 1
  CMR | 8.7 [3.0 to 9.1] | 3.2 [3.1 to 5.5] | 8.9 [8.9 to 8.9]
  MMR: number analyzed (Participants) | 21 | 22 | 17
  MMR | 3.2 [2.7 to 6.0] | 3.2 [2.3 to 6.1] | 3.4 [2.1 to 9.2]

5. Secondary Outcome: Rate of BCR-ABL Undetectable
Description: The BCR-ABL transcript rate was analysed by molecular biology by RQ-PCR at study entry, 3 months, 6 months, 9 months and 12 months.
Time Frame: 12 first months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 24 | 25 | 19
percentage of patients | 29.2 [12.6 to 51.1] | 12.0 [2.5 to 31.2] | 5.3 [0.1 to 26.0]

6. Secondary Outcome: Time to the First BCR-ABL Undetectable
Description: The BCR-ABL transcript rate was analysed by molecular biology by RQ-PCR at study entry, 3 months, 6 months, 9 months and 12 months.
  Time to the first BCR-ABL undetectable was defined by the time from inclusion/randomization and the first CMR.
Time Frame: within 12 months following randomization
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 7 | 3 | 1
Months | 8.7 [3.0 to 9.1] | 3.2 [3.1 to 5.5] | 8.9 [8.9 to 8.9]

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined by the time from de date of inclusion/randomization to the date of death (of any cause).
Time Frame: First 12 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 24 | 25 | 19
Months | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events

8. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined by the time from the date of inclusion and the date of progression.
  Progression was defined as :
  * Death,
  * Passage into the acceleration phase defined by one of the following criteria: % of blood or medullary blasts greater than 15% but less than 30%, blasts plus promyelocytes greater than 30% in the blood or marrow, basophils greater than 20% in the blood, thrombocytopenia less than 100x10^9/L unrelated to treatment, clonal evolution)
  * Passage to the blast transformation phase defined by one of the following criteria: % of blasts of blood or bone marrow greater than 30%, occurrence of extramedullary damage other than histologically proven hepato-splenic.
  * Increase in BCR-ABL transcripts greater than or equal to 2-log compared to the previous values (this increase must be confirmed within 3 months).
Time Frame: First 12 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
Number analyzed (Participants) | 24 | 25 | 19
Months | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: throughout the follow-up of the patient, up to 1 year
Description: All adverse envent (related and unrelated to treatment) were reported.
  All serious adverse envent (related and unrelated to treatment) were reported.
Arm/Group | Imatinib 600 (Randomized Trial) | Imatinib 400 (Randomized Trial) | Imatinib400 (Parallel Cohort)
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/25 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/24 | 4/25 | 0/19
Other Adverse Events (participants affected / at risk) | 24/24 | 12/25 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib 600 (Randomized Trial) (N=24) | Imatinib 400 (Randomized Trial) (N=25) | Imatinib400 (Parallel Cohort) (N=19)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — CARDIAC GENERAL (SOC from CTCAE v3.0)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — CARDIAC GENERAL (SOC from CTCAE v3.0)
Gastrointestinal - Other (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Infection - Other (Specify, __) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — INFECTION (SOC from CTCAE v3.0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — MUSCULOSKELETAL/SOFT TISSUE (SOC from CTCAE v3.0)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — MUSCULOSKELETAL/SOFT TISSUE (SOC from CTCAE v3.0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — PULMONARY/UPPER RESPIRATORY (SOC from CTCAE v3.0)
Renal/Genitourinary - Other (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — RENAL/GENITOURINARY (SOC from CTCAE v3.0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib 600 (Randomized Trial) (N=24) | Imatinib 400 (Randomized Trial) (N=25) | Imatinib400 (Parallel Cohort) (N=19)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) — Immune system disorders (SOC from CTCAE v3.0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) — Immune system disorders (SOC from CTCAE v3.0)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) — Blood and lymphatic system disorders (SOC from CTCAE v3.0)
Leukocytes (total WBC) (Investigations) | 3 (3) | 1 (3) | 1 (2) — Blood and lymphatic system disorders (SOC from CTCAE v3.0)
Lymphopenia (Investigations) | 1 (1) | 1 (3) | 1 (1) — Blood and lymphatic system disorders (SOC from CTCAE v3.0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 (4) | 1 (2) | 1 (1) — Blood and lymphatic system disorders (SOC from CTCAE v3.0)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) — CARDIAC GENERAL (SOC from CTCAE v3.0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) — CARDIAC GENERAL (SOC from CTCAE v3.0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (10) | 3 (4) | 2 (2) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — CONSTITUTIONAL SYMPTOMS (SOC from CTCAE v3.0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1) — DERMATOLOGY/SKIN (SOC from CTCAE v3.0)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — DERMATOLOGY/SKIN (SOC from CTCAE v3.0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) — DERMATOLOGY/SKIN (SOC from CTCAE v3.0)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 0 (0) | 4 (4) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 2 (5) | 1 (1) | 1 (1) — GASTROINTESTINAL (SOC from CTCAE v3.0)
Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — HEMORRHAGE/BLEEDING (SOC from CTCAE v3.0)
Infection - Other (Specify, __) (Infections and infestations) | 6 (8) | 2 (2) | 4 (5) — INFECTION (SOC from CTCAE v3.0)
Edema:head and neck (General disorders) | 3 (6) | 0 (0) | 1 (1) — LYMPHATICS (SOC from CTCAE v3.0)
Edema:limb (General disorders) | 0 (0) | 1 (1) | 1 (1) — LYMPHATICS (SOC from CTCAE v3.0)
Lymphatics - Other (Specify, __) (General disorders) | 0 (0) | 0 (0) | 1 (1) — LYMPHATICS (SOC from CTCAE v3.0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1) — METABOLIC/LABORATORY (SOC from CTCAE v3.0)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — METABOLIC/LABORATORY (SOC from CTCAE v3.0)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 9 (12) | 3 (4) | 2 (2) — MUSCULOSKELETAL/SOFT TISSUE (SOC from CTCAE v3.0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) — NEUROLOGY (SOC from CTCAE v3.0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — OCULAR/VISUAL (SOC from CTCAE v3.0)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2 (2) | 1 (2) | 2 (2) — OCULAR/VISUAL (SOC from CTCAE v3.0)
Watery eye (epiphora, tearing) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — OCULAR/VISUAL (SOC from CTCAE v3.0)
Head/headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) — PAIN (SOC from CTCAE v3.0)
Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) — PAIN (SOC from CTCAE v3.0)
Stomach (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) — PAIN (SOC from CTCAE v3.0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) — PULMONARY/UPPER RESPIRATORY (SOC from CTCAE v3.0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — PULMONARY/UPPER RESPIRATORY (SOC from CTCAE v3.0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — RENAL/GENITOURINARY (SOC from CTCAE v3.0)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) — RENAL/GENITOURINARY (SOC from CTCAE v3.0)
Carotid (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — VASCULAR (SOC from CTCAE v3.0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No